CLINICAL TRIAL: NCT04781088
Title: Phase II Study With Safety Lead-In of Lenvatinib, Pembrolizumab, and Weekly Paclitaxel for Recurrent Endometrial, Epithelial Ovarian, Fallopian Tube and Primary Peritoneal Cancer
Brief Title: Lenvatinib, Pembrolizumab, and Paclitaxel for Treatment of Recurrent Endometrial, Epithelial Ovarian, Fallopian Tube, or Primary Peritoneal Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Floor Backes, MD (Other)
Responsible Party: Sponsor-Investigator, Floor Backes, MD, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-20172; NCI-2021-01256 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2021-02-23; First posted 2021-03-04 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Platinum-Resistant Fallopian Tube Carcinoma; Platinum-Resistant Ovarian Carcinoma; Platinum-Resistant Primary Peritoneal Carcinoma; Recurrent Endometrial Carcinoma; Recurrent Fallopian Tube Carcinoma; Recurrent Ovarian Carcinoma; Recurrent Primary Peritoneal Carcinoma
Keywords: endometrial cancer; ovarian cancer; platinum resistant; phase 2
MeSH Terms: conditions — Endometrial Neoplasms; Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — lenvatinib; Paclitaxel; Taxes; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (paclitaxel, lenvatinib, pembrolizumab) (Experimental): Patients receive paclitaxel IV over 1 hour on days -15 and -8 and lenvatinib PO QD on days -15 to 0. Beginning cycle 1 day 1, patients receive lenvatinib PO QD, pembrolizumab IV over 30 minutes on day 1, and paclitaxel IV over 1 hour on days 1, 8, and 15. Cycles with pembrolizumab repeats every 3 weeks for up to 2 years, and cycles with paclitaxel and lenvatinib repeats every 3 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Lenvatinib; Drug: Paclitaxel; Biological: Pembrolizumab

INTERVENTIONS:
Drug: Lenvatinib — Given PO
  Other Names: E7080; ER-203492-00; Multi-Kinase Inhibitor E7080
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475

SUMMARY:
This phase II clinical trial studies the effect of lenvatinib, pembrolizumab, and paclitaxel in treating patients with endometrial, epithelial ovarian, fallopian tube, or primary peritoneal cancer that has come back (recurrent). While all 3 study drugs are FDA approved, and 2-drug combinations have been studied, the 3- drug combination has not been studied yet. The investigators believe that the addition of pembrolizumab to weekly paclitaxel and lenvatinib (or weekly paclitaxel to pembrolizumab and lenvatinib) is highly effective and safe with manageable side effects in both recurrent endometrial and platinum resistant ovarian cancer. The purpose of this trial is to study how well lenvatinib, pembrolizumab, and weekly paclitaxel work together in women who have recurrent endometrial cancer and/or recurrent platinum resistant ovarian, fallopian tube, and primary peritoneal cancer, and what kind of side effects patients may experience.

DETAILED DESCRIPTION:
PRIAMRY OBJECTIVE:

I. To determine objective antitumor activity (complete and partial response) of lenvatinib, pembrolizumab, and weekly paclitaxel as measured by Response Evaluation Criteria in Solid Tumors (RECIST) criteria in recurrent endometrial and platinum resistant ovarian cancer.

SECONDARY OBJECTIVES:

I. To determine the safety and tolerability weekly paclitaxel, lenvatinib, and pembrolizumab in study patients.

II. To measure the progression free survival in the study population. III. To measure the overall survival in the study population.

EXPLORATORY OBJECTIVE:

I. To explore the baseline tumor genetic and microenvironment parameters predictive of clinical benefit or resistance to the treatment combination and potential mechanisms of resistance.

OUTLINE:

Beginning cycle 1 day 1, patients receive lenvatinib PO daily, pembrolizumab IV on day 1, and paclitaxel IV over 1 hour on days 1, 8, and 15, on a 21 day cycle in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are at least 18 years of age on the day of signing informed consent will be enrolled in this study
* Women with histologically confirmed endometrial cancer, epithelial ovarian cancer, fallopian tube cancer or primary peritoneal cancer (all histological subtypes)
* Patients must have received prior treatment with a platinum containing regimen and may have received 1-3 prior regimens. Hormonal therapy and maintenance therapy (with bevacizumab or PARP inhibitor) does not count towards the number of prior treatments
* Patients with ovarian, fallopian tube or primary peritoneal cancer must be platinum resistant (progression < 6 months after completion of a platinum containing regimen) or not a candidate for further platinum treatment
* Patients with and without mismatch repair deficiency are allowed
* Prior PD-1/PD-L1 inhibitors are allowed as long as this was not the most recent regimen and treatment was not discontinued due to side effects/toxicity. Prior weekly paclitaxel is allowed as long as this was not the most recent regimen and treatment was not discontinued due to side effects/toxicity
* Prior targeted therapy targeting angiogenesis is allowed as long as treatment was not discontinued due to side effects/toxicity
* Have measurable disease based on RECIST 1.1. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions
* A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

  * Not a woman of childbearing potential (WOCBP) as defined OR
  * A WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 4 months (corresponding to time needed to eliminate any study treatment[s] MK and or any active comparator/combination) plus 30 days (a menstruation cycle) after the last dose of study treatment
* The participant (or legally acceptable representative if applicable) provides written informed consent for the trial
* Have provided archival tumor tissue sample or newly obtained core or excisional biopsy of a tumor lesion not previously irradiated. Formalin-fixed, paraffin embedded (FFPE) tissue blocks are preferred to slides. Newly obtained biopsies are preferred to archived tissue.
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
* Absolute neutrophil count (ANC) >= 1500/uL (within 10 days prior to the start of study treatment)
* Platelets >= 100 000/uL (within 10 days prior to the start of study treatment)
* Hemoglobin >= 9.0 g/dL or >= 5.6 mmol/L (within 10 days prior to the start of study treatment)

  * Criteria must be met without erythropoietin dependency and without packed red blood cell (pRBC) transfusion within last 2 weeks
* Creatinine =< 1.5 x upper limit of normal (ULN) OR measured or calculated creatinine clearance (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance [CrCl]) >= 30 mL/min for participant with creatinine levels > 1.5 x institutional ULN (within 10 days prior to the start of study treatment)

  * Creatinine clearance (CrCl) should be calculated per institutional standard
* Total bilirubin =< 1.5 x ULN OR direct bilirubin =< ULN for participants with total bilirubin levels > 1.5 x ULN (within 10 days prior to the start of study treatment)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) =< 2.5 x ULN (=< 5 x ULN for participants with liver metastases) (within 10 days prior to the start of study treatment)
* International normalized ratio (INR) OR prothrombin time (PT) activated partial thromboplastin time (aPTT) =< 1.5 x ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants (within 10 days prior to the start of study treatment)

Exclusion Criteria:

* A women of child birth potential (WOCBP) who has a positive urine pregnancy test within 72 hours prior to registration.
* Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks or 5 half-lives whichever is shorter prior to study entry. Patients may not have received biologics, targeted therapy or immunotherapy for 4 weeks (6 weeks for nitrosoureas or mitomycin C). Hormonal therapy is not considered anti-neoplastic therapy.
* Has received prior radiotherapy within 3 weeks of start of study treatment. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 2-week washout is permitted for palliative radiation (=< 2 weeks of radiotherapy) to non-central nervous system (CNS) disease
* Has received a live vaccine within 30 days prior to the first dose of study drug. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist) are live attenuated vaccines and are not allowed
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug
* Has a known additional malignancy that is progressing or has required active treatment within the past 3 years. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g. breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded
* Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment
* Has severe hypersensitivity (>= grade 3) to pembrolizumab, lenvatinib, or paclitaxel and/or any of its excipients. Note, patients with paclitaxel hypersensitivity are eligible if the if infusion can safely be completed with reduced infusion rates and premedication
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis
* Has a known history of hepatitis B (defined as hepatitis B surface antigen [HBsAg] reactive) or known active hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection. Note: no testing for hepatitis B and hepatitis C is required unless the patient is at risk for, or has symptoms or signs of, hepatitis
* Has a known history of active TB (Bacillus Tuberculosis)
* Known human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with pembrolizumab, lenvatinib and paclitaxel. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated
* Significant cardiovascular disease
* Major surgical procedure (e.g. laparotomy, bowel resection) 4 weeks prior to start of the study drug.
* Neuropathy grade > 1
* Non-healing wound, bone fracture, or skin ulcer
* Active peptic ulcer disease, inflammatory bowel disease, ulcerative colitis, or other gastrointestinal condition with increased risk of perforation; history of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 4 weeks prior to administration of first dose of study drug
* Patients who have a history of a small or large bowel obstruction within 2 weeks of screening or who have and active partial small bowel obstruction or percutaneous endoscopic gastrostomy (PEG)-tube
* Serious/active infection or infection requiring parenteral antibiotics
* Significant arterial or venous thromboembolic disease or vascular disorders within 6 months prior to administration of first dose of study drug, including by not limited to:

  * Cerebrovascular accident (CVA) or transient ischemic attack (TIA)
  * Peripheral ischemia > grade 2 (per Common Terminology Criteria for Adverse Events [CTCAE] version 4.03)
  * Arterial thrombotic event
  * Patients who have a history of deep vein thrombosis or pulmonary embolus < 3 months prior to enrollment must be excluded. However, if patients are on therapeutic anticoagulation, and the deep vein thrombosis (DVT)/pulmonary embolism (PE) has been clinically stable or improved on anticoagulation for > 3 months, patients are eligible.
  * Patients with a history of clotting disorders must be excluded
* Significant bleeding disorders within 6 months prior to administration of first dose of study drug
* Inability to swallow pills, malabsorption syndrome or gastrointestinal disease that severely affects the absorption of study drugs, major resection of the stomach or small bowel, or gastric bypass procedure
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Is pregnant or breastfeeding, or expecting to conceive within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment. Pregnant women are excluded from this study because the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with lenvatinib, breastfeeding should be discontinued if the mother is treated lenvatinib. These potential risks may also apply to other agents used in this study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Objective tumor response | through study completion, an average of 1 year
  Will be assessed by Response Evaluation Criteria in Solid Tumors 1.1. Will be reported as a percentage and will be calculated by the number of patients with a complete or partial response divided by the total number of patients. The percentage of patients with stable disease and progressive disease will be calculated in a similar fashion.

SECONDARY OUTCOMES:
Safety and Toxicity | through study completion, an average of 1 year
  Toxicity as assessed by Common Terminology for Adverse Events version 5.0 will be evaluated descriptively using frequencies and percentages and will be reported using tables. All patients who receive treatment, regardless of eligibility, will be evaluated for toxicity. Toxicities by type and maximum grade over the course of treatment and follow up will be summarized and by date of occurrence.
Progression free survival | through study completion, an average of 1 year
  Time from first therapy to the time of cancer progression, death or lost to follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Floor Backes, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Allegheny Health Network, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu